CLINICAL TRIAL: NCT04021017
Title: PRE-GAIN Bone Health Pilot Study - Physiologic Replacement of EstroGen for Adolescent Females With AnorexIa Nervosa for Bone Health Pilot Study
Brief Title: PRE-GAiN Bone Health Pilot Study
Acronym: PRE-GAiN
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI Workload
Sponsor: University of Saskatchewan (Other)
Collaborators: Jim Pattison Children's Hospital Foundation (Unknown)
Responsible Party: Principal Investigator, Munier Nour, Principal Investigator, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRE-GAiN-01
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Anorexia Nervosa
Keywords: estrogen; anorexia; bone health; bone accrual; IGF-1
MeSH Terms: conditions — Anorexia Nervosa; Anorexia

STUDY DESIGN:
Intervention Model Description: Participants in this study will be randomized 1:1 into 2 groups. One group will receive treatment with a transdermal estrogen patch and the other group will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Participants randomized to the treatment arm will be divided by maturational status:
  * Participants who have had their first period or have a bone age greater than or equal to 14 years will receive PrClimara® 25 (estradiol hemihydrate transdermal system - 25 mcg/day) as a weekly patch, for 24 months.
    o These participants will also receive progesterone (Provera 10 mg tablet) orally every 4 weeks, for 7 days during the second half of the planned menstrual cycle, in order to induce a menstrual period.
  * Participants who have not yet had their first period and have a bone age below 14 years will receive an increasing dose of estrogen. These participants will be initiated on graduated dose of transdermal 17-β estradiol patches:
    * 3.1 mcg/day (1/8 patch) for first six-months,
    * 6.2 mcg/day (1/4 patch) for second six-months,
    * 12.5 mcg/day (1/2 patch) for third six-months, and
    * 25 mcg/day (full patch) for final six-months.
  Interventions: Drug: Estradiol Hemihydrate Transdermal System
- No Treatment (No Intervention): The participants in this group will not receive the estrogen patch nor the oral progesterone.

INTERVENTIONS:
Drug: Estradiol Hemihydrate Transdermal System — Participants who have had their first period or have a bone age greater than or equal to 14 years will receive PrClimara® 25 (estradiol hemihydrate transdermal system - 25 mcg/day) as a weekly patch, for 24 months. Participants who have not yet had their first period and have a bone age below 14 years will receive an increasing dose of estrogen. These participants will be initiated on graduated dose of transdermal 17-β estradiol patches: 3.1 mcg/day (1/8 patch) for first six-months, 6.2 mcg/day (1/4 patch) for second six-months, 12.5 mcg/day (1/2 patch) for third six-months and 25 mcg/day (full patch) for final six-months.
  Other Names: PrClimara® 25
  Arms: Treatment

SUMMARY:
This study will assess the affects of an estradiol hemihydrate transdermal system on bone health in 24 adolescent females aged 12-19 years old with anorexia nervosa. Participants in this study will be randomized 1:1 into 2 groups. One group will receive treatment with a transdermal estrogen patch and the other group will not.

DETAILED DESCRIPTION:
Currently, no therapy exists to improve bone health in females with anorexia nervosa (AN) other than improving body mass. Transdermal estrogen is being investigated as to whether it has benefit to bone health parameters.

While numerous studies have sought to orally replace estrogen in adolescents and women with AN, the replacement therapy suppresses IGF-1, and as a result oral estrogen studies have demonstrated no bone health benefit in AN. However, transdermal physiologic estrogen, due to no first-pass metabolism in the liver, is not IGF-1 suppressive. IGF-1 is known to be hormone that directly affects bone formation and is considered to be osteoanabolic (helps increase bone mass).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 12 - 19 years old
* Meet DSM-5 criteria for Anorexia Nervosa

  o Criteria includes: persistent restriction of energy intake leading to significantly low body weight; either an intense fear of gaining weight or persistent behavior that interferes with weight gain; and a disturbance in the way one's body weight or shape is experienced
* Amenorrhea for at least three months

  * Amenorrhea is a required inclusion criteria as participants with intact menstruation do not meet justification for estrogen replacement (as they are not estrogen deficient)
  * Participants will have been seen and assessed by anorexia clinic physician prior to enrollment to exclude and treat other causes of amenorrhea
* Agree to use a highly effective contraceptive method for the duration of study therapy.

Exclusion Criteria:

* Uncontrolled or chronic medical conditions that may influence bone health (i.e. hyperthyroidism, diabetes mellitus, or celiac disease)
* Use of supraphysiologic corticosteroids for greater than three months
* Pregnancy or attempting pregnancy
* Cigarette smoker
* Known history of a blood clotting disorder (i.e. Factor V Leiden, Protein C Deficiency, etc.)
* Known predisposition to estrogen-related cancers, such as breast or ovarian cancer (e.g. BRCA1)
* Hypersensitivity to this drug or to any ingredient in the formulation or component of the container
* Liver dysfunction or disease as long as liver function tests have failed to return to normal
* Known or suspected estrogen-dependent malignant neoplasia (e.g. endometrial cancer)
* Endometrial hyperplasia
* Known, suspected, or past history of breast cancer
* Undiagnosed abnormal genital bleeding
* Known or suspected pregnancy or lactation
* Active or past history of arterial thromboembolic disease (e.g. stroke, myocardial infarction, coronary heart disease)
* Active or past history of confirmed venous thromboembolism (such as deep vein thrombosis or pulmonary embolism) or active thrombophlebitis
* A high risk of venous or arterial thrombosis, including known thrombophilic disorders
* Partial or complete loss of vision due to ophthalmic vascular disease
* Presence or history of liver tumours (benign or malignant)
* Ongoing use of estrogen containing contraception (oral birth control pill, vaginal ring, patches, depo injections)

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Cortical Wall Thickness | Change from Baseline to Month 24
  Cortical wall thickness as measured by high resolution peripheral quantitative computed tomography (HR-pQCT).

SECONDARY OUTCOMES:
Areal Bone Content | Change from Baseline to Month 24
  Areal bone content as measured by high resolution peripheral quantitative computed tomography (HR-pQCT).
Bone Micro-architectural Parameters | Change from Baseline to Month 24
  Bone micro-architectural parameters as measured by high resolution peripheral quantitative computed tomography (HR-pQCT).
Volumetric Bone Density | Change from Baseline to Month 24
  Volumetric bone density as measured by high resolution peripheral quantitative computed tomography (HR-pQCT).
Bone Strength Estimates | Change from Baseline to Month 24
  Bone strength estimates as measured by high resolution peripheral quantitative computed tomography (HR-pQCT).
Vertebral Fracture Rates | Change from Baseline to Month 24
  Vertebral fracture rates as measured by lateral spine x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Munier Nour, Principal Investigator — Faculty
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No